CLINICAL TRIAL: NCT00004855
Title: A Randomized, Open-Label, Pilot Treatment Trial Evaluating Cellular Dynamics and Immune Restoration in Treatment-Naive HIV-Infected Subjects Receiving Either the Protease Inhibitor LPV/r or the Nucleoside Analogue Reverse Transcriptase Inhibitors d4T/3TC/Abacavir With the Non-Nucleoside Reverse Transcriptase Inhibitor Nevirapine
Brief Title: Effects of Two Anti-HIV Drug Combinations on the Immune Systems of HIV-Infected Patients Who Have Never Received Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5014; 10866 (Registry Identifier: DAIDS ES); ACTG A5014; AACTG A5014; Substudy ACTG AA5036s
Record Dates: First submitted 2000-02-29; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Nevirapine; Stavudine; HIV Protease Inhibitors; Ritonavir; Lamivudine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; ABT 378; abacavir
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; abacavir; Nevirapine; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Abacavir sulfate
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
This study will compare an anti-HIV drug combination of protease inhibitor plus a nonnucleoside reverse transcriptase inhibitor (NNRTI) to one that includes three nucleoside reverse transcriptase inhibitors (NRTIs) plus an NNRTI. NNRTIs, NRTIs, and protease inhibitors are all types of anti-HIV drugs that block the virus in some way.

This study will try to find out if a treatment regimen containing a protease inhibitor plus an NNRTI has a different effect on the rise of CD4 cells compared to a treatment made up of three NRTIs plus an NNRTI. CD4 cells are cells of the immune system that fight infection. This study will also try to see if the combination of drugs used in this study is safe to use in HIV-positive patients.

DETAILED DESCRIPTION:
This study is designed to further define the dynamics and the mechanisms of the CD4 cell rise seen following administration of potent antiretroviral therapy. It will ascertain if treatment regimens containing nucleoside reverse transcriptase inhibitors (NRTIs) with a nonnucleoside reverse transcriptase inhibitor (NNRTI) have different effects on CD4 dynamics than regimens composed of a protease inhibitor with an NNRTI.

Patients are randomized to one of the two treatment arms listed below. They are stratified based on CD4 count and whether they choose to participate in substudy A5036s.

Arm A (protease inhibitor plus NNRTI regimen): At Day 0 (entry), patients begin taking LPV/RTV. At Day 3, patients add NVP, once daily for 2 weeks and then twice daily for the remainder of the study.

Arm B (triple reverse transcriptase inhibitors plus NNRTI regimen): At Day 0 (entry), patients begin taking 3TC plus d4T plus ABC. At Day 3, patients add NVP, once daily for 2 weeks and then twice daily for the remainder of the study.

HIV RNA analysis is performed at Weeks 4 and 5. If the mean is at least 1.0 log10 lower than the baseline HIV RNA, the patient may continue on study treatment. If the mean is not at least 1.0 log10 lower, however, patients are discontinued from the study by no later than Week 8. After 8 weeks of treatment, patients may change antiretroviral medications with permission of the protocol chair or vice chairs. Regular clinical evaluations are conducted. Blood is drawn to determine HIV RNA quantification, absolute CD4 and CD8 counts, immunological evaluations, telomere assays, and part is stored for future testing. Skin testing and return visits for delayed-type hypersensitivity to standard recall antigens are done on three occasions. Patients remain on the study for 48 weeks. Substudy A5036s evaluates viral dynamics during study treatment. Serial plasma samples are collected during the first 24 hours of treatment and at Day 3 and Week 4. Plasma HIV measurements are performed to differentiate between infectious and non-infectious particle production.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 18 years of age or older.
* Are HIV-positive.
* Have a CD4 count of 500 cells/mm3 or less.
* Have a viral load greater than 5,000 and less than 100,000 copies/ml.
* Are willing to use barrier methods of birth control (such as condoms) during the study and for 12 weeks after stopping treatment.
* Will most likely respond well to nevirapine. This is determined by the results of a test.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have ever taken any anti-HIV drugs. (Seven days or less of treatment will be allowed if it was received more than 30 days before study entry.)
* Have pancreatitis (an inflamed pancreas) or hepatitis within 2 weeks of study entry.
* Are pregnant or breast-feeding.
* Actively abuse drugs or alcohol which their doctor feels would interfere with the ability to fulfill study requirements.
* Have taken any medications within 14 days of study entry that would interfere with the study drugs.
* Are receiving or need to receive chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Landay, Study Chair; Michael Lederman, Study Chair
Locations (23):
- United States (23):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Denver Dept of Health and Hosps, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Univ of Texas Galveston, Galveston, Texas

REFERENCES:
- [Derived] Lok JJ, Hunt PW, Collier AC, Benson CA, Witt MD, Luque AE, Deeks SG, Bosch RJ. The impact of age on the prognostic capacity of CD8+ T-cell activation during suppressive antiretroviral therapy. AIDS. 2013 Aug 24;27(13):2101-10. doi: 10.1097/QAD.0b013e32836191b1. PMID 24326304